CLINICAL TRIAL: NCT03135392
Title: Return of Breast Sensation Following Nipple Sparing Mastectomy and Breast Reconstruction With or Without Neurotized Free Tissue Transfer: An Evaluation of Clinical, Sensory, and Quality of Life Outcomes
Brief Title: Sensation After Nipple Sparing Mastectomy and Breast Reconstruction With or Without Neurotized Free Tissue Transfer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research cancelled because of inadequate staffing.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE2117
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Mastectomy; Breast Reconstruction
Keywords: Breast Cancer; sensation recovery; Neurotization
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty; Prostheses and Implants; Nerve Transfer

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study
Who Masked: Participant
Masking Description: Participants who are having implant reconstruction will act as controls for all other breast reconstructions. If the participant is having autologous tissue reconstruction, she will be randomly put into one of the study groups. Neither the study doctor nor the participant can choose the treatment. Assignment is done randomly, like the flip of a coin. If the participant is having only one breast reconstructed, she will be randomly assigned to either receive the nerve reconstruction or not.
  If the participant is having both of her breasts reconstructed, one side will receive the nerve reconstruction and one will not. The participant will not know which group you have been assigned to until the completion of the study or if voluntarily withdraw from the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast Reconstruction with Artificial Implant (Active Comparator): Participants undergoing unilateral reconstruction: patient will serve as internal control with contralateral breast and reconstructed breast will be compared to all other reconstructed breasts. Participants undergoing bilateral reconstruction: reconstructed breasts will be compared to all other reconstructed breasts
  Interventions: Procedure: Breast Reconstruction with Artificial Implant
- Autologous Breast Reconstruction without Neurotization (Active Comparator): Participants undergoing autologous tissue (her own tissue from other areas of the body) reconstruction which do not have their nerves reconstructed during surgery
  Interventions: Procedure: Autologous Breast Reconstruction
- Autologous Breast Reconstruction with Neurotization (Experimental): Participants undergoing autologous tissue (her own tissue from other areas of the body) reconstruction which have a nerve connected (neurotized) during surgery.
  Interventions: Procedure: Autologous Breast Reconstruction; Procedure: Neurotization

INTERVENTIONS:
Procedure: Breast Reconstruction with Artificial Implant — Patients undergo unilateral or bilateral reconstruction of breasts after nipple sparing mastectomy. Breasts are reconstructed with artificial implants
  Arms: Breast Reconstruction with Artificial Implant
Procedure: Autologous Breast Reconstruction — Patients undergo unilateral or bilateral reconstruction of breasts after nipple sparing mastectomy. Breasts are reconstructed with the patient's own tissue
  Arms: Autologous Breast Reconstruction with Neurotization; Autologous Breast Reconstruction without Neurotization
Procedure: Neurotization — Nerve will be reconstructed during autologous breast tissue reconstruction
  Other Names: Nerve Reconstruction
  Arms: Autologous Breast Reconstruction with Neurotization

SUMMARY:
Tissue Expander/Implant Reconstruction: The purpose of this study is to determine how and when nerve sensation to the breast skin returns after mastectomy.

Autologous Tissue Reconstruction: The purpose of this study is to determine whether the tissue being used to reconstruct your breast can provide sensation by using your own nerves. Typically all sensation is lost immediately after this type of surgery and returns to varying degrees. We are hoping to demonstrate that by connecting the two nerves (one from abdomen and one from the chest wall) together, we can attain meaningful sensation in the transferred tissues thereby improving your quality of life following surgery.

DETAILED DESCRIPTION:
To determine the timing and distribution of sensation recovery of breast after mastectomy and breast reconstruction, both with autologous and implant-based reconstruction. Also, to determine the role of innervated free tissue transfer in breast reconstruction.

Specific Aims

1. Determine the timing and degree of return of breast in women who underwent mastectomy with autologous tissue or with implant based reconstruction.
2. Determine sensation following neurotized free flap reconstruction
3. Determine whether neurotization has an impact on quality of life measures post operatively

Study Design Patients will be enrolled prospectively in this data collection study in which they will receive the standard of care for breast cancer resection and oncologically safe and accepted means of breast reconstruction with tissue expander and/or prosthetic implants. Patients will receive additional, non-invasive sensory testing, performed at standard follow up intervals in clinic by their reconstructive team. All patients participating in the study will be consented for enrollment at the pre-operative visit by either the surgeon or physician assistant. As this is a prospective study, all women fitting inclusion criteria over a 6-month minimal, but projected goal 12-month period will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral or bilateral skin sparing mastectomy for breast cancer
* Patient must have one of the following reconstructions in planned:

  * Immediate tissue expander placement
  * Immediate implant placement
  * Immediate autologous breast reconstruction
* All patients participating in the study must be willing to be consented for enrollment at the pre-operative visit.

Exclusion Criteria:

* Pre-operative radiation therapy
* Any pre-excising
* Patients with absent or prior damaged nipple areola-complex (NAC) on the "non-surgical breast"

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Composite measure of sensation | Up to 24 months after surgery
  Differences of at least 20% comparing control to experimental breasts would be clinically meaningful. Composite measure will be calculated by combining the follow binomial factors: detection of temperature difference (feeling hot and cold), detection of sharp versus dull pressure, detection of vibration, discerning point pressure

SECONDARY OUTCOMES:
Quality of Life as measured by a 19-question survey regarding sensation and appearance of breast. | Up to 24 months after surgery
  A total of 19 Likert scale questions will be given to participants in the pre- and post-Surgical Sensation Questionnaire regarding sensation and appearance of breast before and after reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Moreira, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States